CLINICAL TRIAL: NCT04736199
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of Darolutamide in Addition to Androgen Deprivation Therapy (ADT) Versus Placebo Plus ADT in Men With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Brief Title: Darolutamide in Addition to ADT Versus ADT in Metastatic Hormone-sensitive Prostate Cancer
Acronym: ARANOTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21140; 2022-502244-12-00 (Other: CTIS (EU)); 2020-003093-48 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: Metastatic hormone-sensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darolutamide+ADT (Experimental): Participants will receive darolutamide 600 mg (2 tablets of 300 mg) twice daily with food and ADT of investigator's choice as standard therapy
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788); Other: Androgen deprivation therapy (ADT)
- Placebo+ADT (Placebo Comparator): Participants will receive placebo twice daily with food and ADT of investigator's choice as standard therapy
  Interventions: Drug: Placebo; Other: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — Coated tablet, oral administration
  Arms: Darolutamide+ADT
Drug: Placebo — Coated tablet matching Darolutamide in appearance, oral administration
  Arms: Placebo+ADT
Other: Androgen deprivation therapy (ADT) — Luteinizing hormone-releasing hormone (LHRH) agonist/antagonists or orchiectomy

SUMMARY:
The purpose of the study is to assess the efficacy and safety of darolutamide in combination with standard androgen deprivation therapy (ADT) in patients with metastatic hormone sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate
* Metastatic disease
* Started ADT (LHRH agonist/antagonist or orchiectomy) with or without first generation anti-androgen, but not earlier than 12 weeks before randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1 or 2
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior treatment with: LHRH agonist/antagonists except neoadjuvant and /or adjuvant therapy; Second-generation androgen receptor (AR) inhibitors such as enzalutamide, darolutamide, apalutamide or other investigational AR inhibitors; Cytochrome P17 enzyme inhibitor such as abiraterone acetate or oral ketoconazole as anti-cancer treatment for prostate cancer; Chemotherapy including docetaxel or immunotherapy for prostate cancer; Use of systemic corticosteroid with dose greater than the equivalent 10 mg of prednisone/day within 28 days prior to randomization; Radiopharmaceuticals; Any other anti-cancer treatment for prostate cancer, excluding local therapies and ADT.
* Treatment with radiotherapy within 2 weeks before randomization
* Contraindication to iodinated CT and gadolinium chelate MRI intravenous contrast agent(s)
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV)
* Uncontrolled hypertension as indicated by a resting systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite medical management
* A gastrointestinal (GI) disorder or procedure which is expected to interfere significantly with absorption of study drug
* Any prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) within 5 years prior to randomization
* Inability to swallow oral medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (131):
- Australia (6):
  - Nepean Hospital, Kingswood, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Macquarie University Hospital - Oncology Department, Sydney, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
  - Peninsula Oncology Centre, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
- Brazil (16):
  - Assistência Multidisciplinar em Oncologia (AMO), Salvador, Estado de Bahia
  - Hosp. Araujo Jorge da Associação de Combate ao Câncer, Goiânia, Goiás
  - Hospital da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Cetus Oncologia Hospital Dia, Belo Horizonte, Minas Gerais
  - Liga Paranaense de Combate ao Cancer-Hosp Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer | Centro de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Unidade de Pesquisas Clinicas em Oncologia, Pelotas, Rio Grande do Sul
  - Santa Casa de Porto Alegre | Hospital Sao Francisco - Centro Medico Pesquisa Clinica Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - FZ Pesquisa e Servicos em Cardiologia | Porto Alegre, Brazil, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos/SP, São Paulo
  - Hospital de Base | Funfarme - Centro Integrado de Pesquisa - Cardiologia, São José do Rio Preto, São Paulo
  - Urobrasil, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Inst. de Assistência Médica ao Sérvidor Público Estadual, São Paulo, São Paulo
  - Instituto COI de Educação e Pesquisa, Rio de Janeiro
- Canada (2):
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal (CRCHUM), Montreal, Quebec
- Chile (7):
  - Centro de Investigación Clínica del Sur, Temuco, Región de la Araucanía
  - OncoCentro, Viña del Mar, Región de Valparaíso
  - Centro de Estudios Clínicos SAGA SpA, Providencia, Santiago Metropolitan
  - Fundación Arturo López Perez, Santiago
  - Oncovida, Santiago
  - Hospital Clínico de la Pontificia Univ. Católica de Chile, Santiago
  - UROMED, Santiago
- China (25):
  - Anhui Provincial Hospital, Hefei City, Anhui Province, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People Hospital, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Zhongnan hospital ,Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Nantong tumor hospital, Nantong, Jiangsu
  - The 2nd Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - 1st Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shengyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - SichuanAcademyofMedicalSciences&SichuanProvincialPeople'sHos, Chengdu, Sichuan
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - The 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
- India (23):
  - Mahatma Gandhi Cancer Hospital & Research Institute, Visakhapatnam, Andhra Pradesh
  - The Gujarat Cancer & Research Institute, Ahmedabad, Gujarat
  - HCG Cancer Centre - Ahmedabad, Ahmedabad, Gujarat
  - Cancer Care Clinic - Vadodara, Vadodara, Gujarat
  - K.L.E.S. Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - Healthcare Global Enterprises Ltd, Bengaluru, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Marathwada Regional Cancer Centre and Research Institute, Aurangabad, Maharashtra
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Sparsh Hospital & Critical Care, Bhubaneswar, Odisha
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Jawaharlal Institute Of Postgraduate Medical Education and R, Gorimedu, Puducherry
  - Christian Medical Center & Hospital, Ludhiana, Punjab
  - Sawami Man Singh (SMS) Medical College & Attached Hospitals, Jaipur, Rajasthan
  - Apollo Speciality Hospitals, Madurai, Tamil Nadu
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Tata Medical Center, Kolkata
  - Apex Wellness Hospital, Nashik
  - Rajiv Gandhi Cancer Institute & Research Centre, New Delhi
- Latvia (5):
  - Daugavpils Regional Hospital, Daugavpils
  - RAKUS Hospital Gailezers, Riga
  - URO Ltd., Riga
  - P. Stradins Clinical University Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (4):
  - The Hospital of Lithuanian University of Health SciencesLUHS, Kaunas
  - PI Klaipedos University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- New Zealand (3):
  - Canterbury Urology Research Trust, Christchurch, Canterbury
  - Waikato Hospital, Hamilton
  - Tauranga Urology Research Limited, Tauranga
- Peru (4):
  - Aliada, San Isidro, Lima region
  - Hospital Guillermo Almenara Irigoyen, Santiago de Surco, Lima region
  - Hospital Militar Luis Arias Schreiber, Lima
  - Clínica El Golf, Lima
- Russia (17):
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - Ltd "EVIMED", Chelyabinsk
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Republican Clinical Oncology Dispensary Kazan, Kazan'
  - Research Centre of X-ray and Radiology, Moscow
  - Volga District Med Center FMBA, Nizhny Novgorod
  - LLC Reafan, Novosibirsk
  - Medical Center "Avicenna", Novosibirsk
  - Clinical Oncological Dispensary of Omsk Region, Omsk
  - AV Medical Group, Saint Petersburg
  - Russian Scientific Radiology and Surgery Technologies Center, Saint Petersburg
  - Scientific Research Instutute of Oncology n.a. N.N. Petrov, Saint Petersburg
  - Multi-Field Clinical Medical Center "Medical City", Tyumen
  - Republican Clinical Oncology Dispensary, Ufa
  - Vologda Regional Hospital, Vologda
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- South Africa (4):
  - Cancercare Langenhoven, Port Elizabeth, Eastern Cape
  - East Rand Medical Research Unit, Johannesburg, Gauteng
  - University of Pretoria, Clinical Research Unit, Pretoria, Gauteng
  - Cape Town Oncology Trials, Cape Town
- Spain (6):
  - Hospital Universitario Fundacion Alcorcon | Urologia, Alcorcón, Madrid
  - Fundacio Puigvert | Urologia, Barcelona
  - Parc Tauli Hospital Universitari | Oncologia, Barcelona
  - Hospital San Pedro De Alcantara | Oncologia, Cáceres
  - Hospital Universitario Virgen De La Victoria | Urologia, Málaga
  - Hospital Universitario Virgen Del Rocio S.L. | Urologia, Seville
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Changhua Christian Hospital, Changhua
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Ukraine (4):
  - CNE "Clinical Center of Oncology, Hematology, Transplantology and Palliative Care of the Cherkasy Regional Council", Cherkasy
  - City Dnipropetrovsk Multi- field Clinical Hosp. 4 DSMA, Dnipro
  - Kyiv City Hospital #3 - Department of Urology, Kyiv
  - Kyiv Regional Oncological Dispensary, Kyiv

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Saad F, Vjaters E, Shore N, Olmos D, Xing N, Pereira de Santana Gomes AJ, Cesar de Andrade Mota A, Salman P, Jievaltas M, Ulys A, Jakubovskis M, Kopyltsov E, Han W, Nevalaita L, Testa I, Le Berre MA, Kuss I, Haresh KP; ARANOTE Study Investigators. Darolutamide in Combination With Androgen-Deprivation Therapy in Patients With Metastatic Hormone-Sensitive Prostate Cancer From the Phase III ARANOTE Trial. J Clin Oncol. 2024 Dec 20;42(36):4271-4281. doi: 10.1200/JCO-24-01798. Epub 2024 Sep 16. PMID 39279580
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 133 centers in Europe/Rest of the world (ROW), Asia, and Latin America between 23-Feb-2021 (first participant first visit) and 07-Jun-2024 (primary completion date). Study is still ongoing.
Pre-assignment Details: In total 889 participants were screened in the study and 202 participants were screen failures. An additional 18 participants prematurely discontinued screening. A total of 669 participants were randomized (446 to the darolutamide arm and 223 to the placebo arm).
Groups:
- Darolutamide+ADT: Participants received darolutamide (BAY1841788) 600 mg (2 tablets of 300 mg) twice daily with food and androgen deprivation therapy (ADT) of investigator's choice as standard therapy.
- Placebo+ADT: Participants received matching placebo twice daily with food and androgen deprivation therapy (ADT) of investigator's choice as standard therapy.
Period: Overall Study
Arm/Group | Darolutamide+ADT | Placebo+ADT
Started | 446 | 223
Treated | 443 | 223
Completed | 0 | 0
Not Completed | 446 | 223
Not completed — Adverse Event | 28 | 22
Not completed — Death | 9 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 5 | 9
Not completed — Withdrawal by Subject | 21 | 9
Not completed — Progressive disease | 120 | 101
Not completed — Subject decision | 13 | 13
Not completed — Required study drug interruption longer than allowed per protocol | 2 | 0
Not completed — Additional primary malignancy | 1 | 0
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Other reason | 0 | 1
Not completed — Ongoing with study drug | 240 | 63
Not completed — Study drug never administered | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darolutamide+ADT | Placebo+ADT | Total
Number analyzed (Participants) | 446 | 223 | 669
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (8.8) | 69.2 (8.9) | 69.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 446 | 223 | 669
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104 | 58 | 162
  Not Hispanic or Latino | 334 | 157 | 491
  Unknown or Not Reported | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 251 | 125 | 376
  Black or African American | 41 | 24 | 65
  Asian | 144 | 65 | 209
  Other | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Radiological Progression-free Survival (rPFS) Assessed by Central Review
Description: rPFS used conventional imaging method (99mTc-phosphonate bone scan, CT/MRI scan). rPFS was defined as the time from the date of randomization to the date of progressive disease in malignant soft tissue lesions, progressive disease in malignant bone lesions, or death due to any cause, whichever occurs first. Malignant soft tissue lesions were assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and malignant bone lesions were assessed by Prostate Cancer Clinical Trials Working Group (PCWG3) criteria.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | 25.0 [19.0 to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; Analyzed with log-rank test and Cox regression proportional hazard model, stratified by the same factor as used for randomization visceral disease (present versus absent), prior local therapy (Yes versus No); Test type: Superiority; p < 0.0001, Log Rank — One-sided; Hazard Ratio (HR) = 0.541, 95% CI 2-sided [0.413 to 0.707]

2. Secondary Outcome: Overall Survival (OS)
Description: Time from the date of randomization to the date of death from any cause.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | NA [33.8 to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1007, Log Rank — One-sided; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.591 to 1.118] — significance level of 0.0185 (one-sided)

3. Secondary Outcome: Time to Castration-Resistant Prostate Cancer (CRPC)
Description: Time from the date of randomization to the date of first castration resistant event (radiological progression, Prostate-specific antigen (PSA) progression or symptomatic skeletal events, whichever occurs first).
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | 13.8 [12.0 to 16.8]
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.404, 95% CI 2-sided [0.321 to 0.508]

4. Secondary Outcome: Time to Initiation of Subsequent Anti-cancer Therapy
Description: Time from the date of randomization to initiation of first subsequent anti-cancer therapy for prostate cancer.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | NA [27.7 to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.401, 95% CI 2-sided [0.288 to 0.558]

5. Secondary Outcome: Time to PSA Progression
Description: Time from the date of randomization to the date of first prostate-specific antigen (PSA) progression. PSA progression with serum testosterone being at castrate level <0.50 ng/mL, is defined as a ≥25% increase above the nadir (lowest at or after baseline) value and an increase in absolute value of ≥2 ng/mL above nadir, and is at least 12 weeks from randomization date, which is confirmed by a second value 3 or more weeks later. All PSA values between the initial assessment meeting the PSA progression criteria and confirmation assessment must be ≥2 ng/mL and ≥25% increase above nadir, serum testosterone at castrate levels <0.50 ng/mL is requested at initial assessment.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | 16.8 [13.9 to 20.1]
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.306, 95% CI 2-sided [0.231 to 0.405]

6. Secondary Outcome: PSA Undetectable Rates (<0.2 ng/mL)
Description: Percentage of subjects with detectable PSA values of ≥0.2 ng/mL at baseline which became undetectable with any PSA values <0.2 ng/mL during the period between randomization and 30 days after last dose of study drug or start of new anti-cancer therapy whichever occurred earliest, based on the subjects had detectable PSA value at baseline.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Participants with detectable PSA values ≥0.2 ng/mL at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 425 | 211
Percentage of participants | 62.6 [57.8 to 67.2] | 18.5 [13.5 to 24.4]
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Other; Rate difference = 44.3, 95% CI 2-sided [37.4 to 51.2]

7. Secondary Outcome: Time to Pain Progression
Description: Pain progression was assessed by Question 3 (Q3) of the BPI-SF questionnaire related to the worst pain in the last 24 hours (worst pain subscale [WPS]) taken as an average for post baseline score, or initiation of short or long-acting opioids for malignant disease for ≥7 consecutive days after randomization. Pain progression was defined as: (1) for asymptomatic subjects with WPS=0 at baseline, an increase of 2 or more points in the WPS score from nadir observed at 2 consecutive evaluations ≥4 weeks apart, or initiation of short- or long-acting opioid use for malignant disease for ≥7 consecutive days after randomization; (2) for symptomatic subjects with WPS >0 at baseline, an increase of 2 or more points in the WPS score from nadir observed at 2 consecutive evaluations ≥4 weeks apart and a WPS ≥5, or initiation of short- or long-acting opioid use for malignant disease for ≥7 consecutive days after randomization.
Time Frame: From randomization to the date when 222 rPFS events were observed, approximately 36 months
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 446 | 223
Months | NA [NA to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events. | 29.9 [29.7 to NA] — NA signifies that value cannot be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Darolutamide+ADT vs Placebo+ADT; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.721, 95% CI 2-sided [0.544 to 0.957]

8. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, after providing written IC for participation in the study, may or may not be temporally associated with the use of study drug, whether or not considered related to the study drug. Treatment-emergent AE (TEAE) is defined as any event arising or worsening after the first dose of study drug until 30 days after the last dose of study drug.
Time Frame: From start of study drug administration until 30 days after the last administration
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Darolutamide+ADT | Placebo+ADT
Number analyzed (Participants) | 445 | 221
Participants
  Any TEAE | 405 | 199
  Any TESAE | 105 | 52
  Any study drug-related TEAE | 144 | 64

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last administration. All-cause mortality death events at any time during the study, up to cut-off date for the primary completion analysis 07 JUN 2024 (approximately 39 months).
Groups:
- Darolutamide + ADT: Participants received darolutamide (BAY1841788) 600 mg (2 tablets of 300 mg) twice daily with food and androgen deprivation therapy (ADT) of investigator's choice as standard therapy.
- Placebo + ADT: Participants received matching placebo twice daily with food and androgen deprivation therapy (ADT) of investigator's choice as standard therapy.
Arm/Group | Darolutamide + ADT | Placebo + ADT
All-Cause Mortality (participants affected / at risk) | 105/445 | 61/221
Serious Adverse Events (participants affected / at risk) | 105/445 | 52/221
Other Adverse Events (participants affected / at risk) | 321/445 | 149/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide + ADT (N=445) | Placebo + ADT (N=221)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (2) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (10) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 2 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 5 (6) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary calculus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostate ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Device expulsion (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide + ADT (N=445) | Placebo + ADT (N=221)
Anaemia (Blood and lymphatic system disorders) | 89 (101) | 37 (42)
Constipation (Gastrointestinal disorders) | 42 (43) | 16 (17)
Fatigue (General disorders) | 25 (26) | 18 (19)
Urinary tract infection (Infections and infestations) | 48 (63) | 17 (27)
COVID-19 (Infections and infestations) | 32 (35) | 14 (15)
Alanine aminotransferase increased (Investigations) | 39 (45) | 18 (18)
Aspartate aminotransferase increased (Investigations) | 42 (47) | 17 (18)
Blood creatinine increased (Investigations) | 21 (22) | 15 (20)
Weight increased (Investigations) | 33 (39) | 17 (19)
Blood alkaline phosphatase increased (Investigations) | 30 (33) | 13 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 27 (34) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 (63) | 25 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (54) | 22 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 31 (34) | 26 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (44) | 18 (23)
Headache (Nervous system disorders) | 18 (23) | 14 (15)
Insomnia (Psychiatric disorders) | 28 (30) | 6 (6)
Hypertension (Vascular disorders) | 38 (41) | 19 (21)
Hot flush (Vascular disorders) | 41 (43) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04736199/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04736199/SAP_001.pdf